CLINICAL TRIAL: NCT05003011
Title: Correlation of Hemodynamics Via Pulmonary Artery Catherization and the Cardiospire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Respirix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD-02-1511
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Hemodynamic Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Cardiospire — Non-invasive hemodynamic monitoring

SUMMARY:
This study is designed as an observational study to collect Cardiospire cardiogenic oscillation signal (COS) and CO output parameters from the Pulmonary Artery Catheter in intubated patients.

DETAILED DESCRIPTION:
Respirix has developed a non-invasive hemodynamic monitoring device called the Cardiospire. The Cardiospire detects minor, cyclic waveforms caused by Cardiogenic Oscillations (COS) and uses features of the COS waveform to provide information about hemodynamics.

This study is designed as an observational study to collect paired readings of the Cardiospire cardiogenic oscillation signal (COS) and the ground truth CO output parameters, including Pulmonary Artery Pressure diastolic (PAPd), systolic (PAPs), Stroke Volume (SV), and Cardiac Output (CO) from the Pulmonary Artery Catheter in intubated patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Intubated
* Pulmonary artery catheter
* Patient or patient's legally authorized representative is able to provide informed consent

Exclusion Criteria:

* Subjects who, at the principal investigator's determination, would not be appropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated patients in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Repeatable Data Verification | 3 months
  First 10 patient Cardiospire data will be processed and analyzed to determine if deemed repeatable for cardiogenic oscillations (COS).
Correlation and Validation of data | 1.5 years
  Collected Cardiospire data from next 150 patients will be analyzed in comparison to PAC data for correlation and validation purposes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States